CLINICAL TRIAL: NCT04473274
Title: GlitazOne Treatment for Coronavirus HypoxiA, a Safety and Tolerability Open Label With Matching Cohort Pilot Study
Acronym: GOTCHA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samaritan Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-042
Record Dates: First submitted 2020-06-22; First posted 2020-07-16 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus Infection; Diabetes
Keywords: COVID19; Diabetes; COVID-19; Coronavirus
MeSH Terms: conditions — Coronavirus Infections; Diabetes Mellitus; COVID-19 | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Matching cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone group (Experimental): Participants will receive pioglitazone 15mg to 30mg daily oral or enteral during hospitalization for up to 30 days in addition to standard of care
  Interventions: Drug: Pioglitazone
- Matching cohort group (No Intervention): Participants will standard of care

INTERVENTIONS:
Drug: Pioglitazone — Receive pioglitazone 15mg - 30mg daily
  Arms: Pioglitazone group

SUMMARY:
Pioglitazone is an approved anti-hyperglycemic medication and is thought to have anti-inflammatory properties. This study seeks to gather safety and tolerability data related to pioglitazone when given to patients who require hospital admission for confirmed positive COVID-19 infections with elevated blood sugar levels as compared to patients who did not receive pioglitazone during their hospitalization for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Laboratory confirmed COVID-19 requiring hospitalization
* A1c greater than 5.6% as measured in the last 30 days
* Women of child-bearing potential who agree to use highly effective method of contraception (defined as either abstinence, condom, diaphragm, and/or oral or injected hormonal contraception) during dosing and for 30 days after last dose
* MRSA PCR screen negative

Exclusion Criteria:

* Pregnancy or nursing
* Congestive Heart Failure all classes (NYHA Class I, II, III or IV)
* Liver enzyme ALT greater than 2.5 times upper limit of normal
* End stage renal disease
* Hypersensitivity or allergy to a TZD (thiazolidinedione)
* Active bladder cancer
* Currently taking a beta blocker, a CYP2C8 inhibitor or inducer such as gemfibrozil or rifampin, a TZD
* Other current or historical illness that in the opinion of the investigator at attending provider would interfere with the subject's ability to complete the study or make it not in the best interest of the subject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Adverse events outcomes without attribution | Baseline, until 30 days after last dose
  Number and type of adverse events
Adverse events attributable | Baseline, until 30 days after last dose
  Number and type of adverse events

SECONDARY OUTCOMES:
Clinical improvement | Baseline, until 30 days after last dose
  Disease severity as measured by 7 point ordinal scale
Levels of treatment | Baseline, until 30 days after last dose
  Type of oxygen support treatment
d-Dimer | Baseline, until 30 days after last dose
  Change from Baseline of d-Dimer
C Reactive Protein | Baseline, until 30 days after last dose
  Change from Baseline of CRP
Ferritin | Baseline, until 30 days after last dose
  Change from Baseline of Ferritin
Lactate dehydrogenase | Baseline, until 30 days after last dose
  Change from Baseline of Lactate dehydrogenase
A1c | Baseline, until 30 days after last dose
  Change from Baseline of A1c

CONTACTS AND LOCATIONS:
Overall Officials: Brian Delmonaco, MD, Principal Investigator — Samaritan Health Services
Locations (1):
- Good Samaritan Hospital Corvallis, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No